CLINICAL TRIAL: NCT06973668
Title: A Randomized Study to Compare Post-transplant Cyclophosphamide, Sirolimus, Ruxolitinib and Post-transplant Cyclophosphamide, Sirolimus, Mycophenolate Mofetil to Prevent Graft Versus Host Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1940; NCI-2025-03239 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: AML
MeSH Terms: interventions — Mycophenolic Acid; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 01A:Treatment With Post-Transplant Cyclophosphamide (PTCy), Sirolimus and MMF (Experimental): 15 mg/kg/dose (max: 1,000mg/dose) IV/PO three times daily
  Interventions: Drug: Mycophenolate Mofetil
- 01B:Treatment With Post-Transplant Cyclophosphamide (PTCy),Sirolimus and Ruxolitinib (Experimental): 5 mg PO every 12 hours
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 15 mg/kg/dose (max: 1,000mg/dose) IV/PO three times daily
  Arms: 01A:Treatment With Post-Transplant Cyclophosphamide (PTCy), Sirolimus and MMF
Drug: Ruxolitinib — 5 mg PO every 12 hours
  Other Names: Jakafi®
  Arms: 01B:Treatment With Post-Transplant Cyclophosphamide (PTCy),Sirolimus and Ruxolitinib

SUMMARY:
The goal of this clinical research study is to compare the effects of these drug combinations (cyclophosphamide, sirolimus, and MMF vs cyclophosphamide, sirolimus, and ruxolitinib) on the prevention of GVHD after a stem cell transplant.

DETAILED DESCRIPTION:
Primary Objective:

To compare Grade 2-4 acute graft versus host disease-free survival (GFS) between the MMF and Ruxolitinib arms

Secondary Objectives:

To compare the following between treatment arms:

1. Grade 3-5 adverse event of this regimen as per CTCAE v5.0 criteria.
2. Graft versus host disease-free, relapse-free survival (GRFS)
3. Time to neutrophil and platelet engraftment
4. Incidence of acute and chronic GVHD
5. Relapse incidence
6. Non relapse mortality
7. Overall survival
8. Progression-free survival
9. Chimerism
10. Immunosuppression cessation time
11. Rate of graft failure

Exploratory Objective:

To conduct mechanistic studies to compare immune recovery between arms and correlate these with disease control and GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 and < 75 years are eligible if they have one of the following diseases.

   1. Acute Myeloid Leukemia
   2. Myelodysplastic syndrome
   3. Chronic myelomonocytic leukemia
2. Available HLA-identical or haploidentical related donor or a 7/8 or 8/8 HLA matched unrelated donor.
3. Peripheral blood stem cells as a graft source
4. Subject must voluntarily sign an informed consent.
5. Adequate organ function per local laboratory reference range as follows: - Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0X ULN - Total Bilirubin <1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of nonhepatic origin) - Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 40 mL/min/1.73 m2 (as reported in epic using 2021 CKD-EPI creatinine equation)

   * DLCO corrected for Hgb, if applicable) ≥ 50% of predicted
   * Ejection Fraction ≥ 50%
   * The effects on the developing human fetus are unknown. For this reason and as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

     * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
     * History of hysterectomy or bilateral salpingo-oophorectomy.
     * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
     * History of bilateral tubal ligation or another surgical sterilization procedure.

Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study agent administration.

Exclusion Criteria:

1. Subject is known to be positive for HIV.
2. Subject has acute promyelocytic leukemia.
3. Subject has known active CNS involvement with AML.
4. Hematopoietic Cell Transplantation Comorbidity Index (HCT-CI) score of >5
5. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
   2. Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or subjects with positive anti-HBc antibody but negative Hep B DNA may participate.
6. Cardiac history of CHF requiring treatment or Ejection Fraction < 50% or unstable angina or MI within 1 year of study entry
7. Major adverse cardiac events such as MI/stroke and pulmonary embolism (PE)/deep vein thrombosis (DVT) within 6 months. Recent history of Central line-associated DVT may be allowed after discussion with PI.
8. Current and/or history of active TB
9. White Blood Cell count > 25 X 109 /L.
10. Pregnant women are excluded from this study because the study agent has unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with the study agent. These potential risks may also apply to other agents used in this study.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, MBA,MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org